CLINICAL TRIAL: NCT00824850
Title: Characterization of the Prevnar Infant Long-term Immune Response vs a Prevnar Naive Cohort
Brief Title: Study Evaluating Prevnar Infant Long-term Immune Response Versus Prevnar Naive Cohort
Acronym: PILOT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 6096A1-3016; B1851014
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Results first posted 2011-11-11 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-10

CONDITIONS: Pneumococcal Conjugate Vaccine
Keywords: Single site; single dose; Participated in Wyeth D118-P8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Subjects received Prevnar in study D118-P8
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- 2 (Experimental): Subjects received MnCC in study D118-P8
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine — single injection, single dose, single site, 0.5 mL per dose.
  Other Names: 13vPnC
  Arms: 1
Biological: 13-valent Pneumococcal Conjugate Vaccine — single injection, single dose, single site, 0.5 mL per dose.
  Other Names: 13vPnC
  Arms: 2

SUMMARY:
The purpose of this study is to assess the "late" immune response to further doses of pneumococcal conjugate vaccine more than 10 years after primary immunization with Prevnar (7vPnC) in infancy, as compared with individuals who did not receive Prevnar in infancy (the Prevnar naive cohort which received MnCC). The study will take place at a single study center. Study participants must have participated previously in a specific Wyeth Prevnar study (Study D118-P8) and must still be enrolled in the Northern California Kaiser Permanente (NCKP) health plan.

ELIGIBILITY:
Inclusion Criteria:

* Fully vaccinated per-protocol (4 doses of vaccine given at 2, 4, 6, and 12-15 months of age) subjects enrolled in the Prevnar arm of Study D118-P8, OR
* Fully vaccinated per-protocol subjects from the control arm of the same study that did not receive Prevnar after the close of Study D118-P8, or at any time following the study, AND
* Still enrolled in NCKP health plan.
* Subjects included in either group above must be in good health as determined by medical history, physical examination, and clinical judgment.

Exclusion Criteria:

* Previous receipt of pneumococcal polysaccharide vaccine.
* History of documented recurrent pneumococcal otitis media or any occurence of pneumonia within past 12 months
* History of documented invasive pneumococcal disease (defined as a positive culture of S. pneumoniae from a normally sterile body site).
* Known or suspected disease or dysfunction of the immune system, including:
* HIV infection
* Malignancy
* Receipt of immunosuppressive therapy
* Sickle cell hemoglobinopathy
* Concomitant vaccination during the study period.
* Known hypersensitivity to any component of Prevnar.
* Any major illness/condition that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in and completion of, the study, or could preclude the evaluation of the subject's response.
* Receipt of immune globulin within the past 3 months.
* Positive pregnancy test for menarchal female subjects.
* Females who are breastfeeding.
* For control subjects, previous receipt of Prevnar at any time.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Hayward, California
  - Pfizer Investigational Site, San Jose, California

REFERENCES:
- [Derived] Klein NP, Ensor K, Jouve S, Northington R, Moscariello M, McGovern PC. Long-term immune responses to pneumococcal conjugate vaccines in children previously vaccinated with 7-valent pneumococcal conjugate vaccine. Pediatr Infect Dis J. 2013 Sep;32(9):990-7. doi: 10.1097/INF.0b013e3182959f34. PMID 24008739
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-3016&StudyName=Study%20Evaluating%20Prevnar%20Infant%20Long-term%20Immune%20Response%20versus%20Prevnar%20Naive%20Cohort

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were previously enrolled in Prevnar protocol D118-P8 (study duration 1995 to 1998) and were randomized to receive either 7-valent pneumococcal conjugate vaccine or meningococcal C conjugate vaccine in that study.
Groups:
- 7vPnC / 13vPnC: 13vPnC administered as a single 0.5 mL dose IM. Participants had previously received 7vPnC in study D118-P8.
- MnCC / 13vPnC: 13vPnC administered as a single 0.5 mL dose IM. Participants had previously received MnCC in study D118-P8.
Period: Overall Study
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Started | 38 | 37
Received Vaccination 13vPnC | 38 | 36
Completed | 38 | 36
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC | Total
Number analyzed (Participants) | 38 | 37 | 75
Age Continuous [Mean (Standard Deviation); unit: years] | 12.6 (1.1) | 13.1 (0.9) | 12.8 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Pneumococcal IgG Antibody Concentration ≥0.35 Mcg/mL for the 13 Serotypes for 7vPnC / 13vPnC in Comparison to MnCC / 13vPnC After Vaccination (Visit 5)
Description: Percentage of participants achieving predefined IgG antibody threshold ≥0.35 micrograms per milliliter (Mcg/mL) for the 13 pneumococcal serotypes (7vPnC serotypes 4, 6B, 9V, 14, 18C, 19F, 23F and additional serotypes 1, 3, 5, 6A, 7F, and 19A) along with the exact, 2-sided 95% confidence intervals (CIs) based on the observed percentage of participants.
Time Frame: Day 28 (Visit 5)
Population: Evaluable Immunogenicity population: eligible participants based on all inclusion and exclusion criteria, had a baseline blood sample collection performed (Visit 1), received 1 dose of 13vPnC, and had Visit 5 blood sample collection performed, and at least 1 valid and determinate assay result at Visit 1 and also at Visit 5.
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Number analyzed (Participants) | 38 | 35
observed percentage of participants
  7vPnC serotype 4 | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  7vPnC serotype 6B | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  7vPnC serotype 9V | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  7vPnC serotype 14 | 100.0 [90.7 to 100.0] | 97.1 [85.1 to 99.9]
  7vPnC serotype 18C | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  7vPnC serotype 19F | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  7vPnC serotype 23F | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 1 | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 3 | 94.7 [82.3 to 99.4] | 97.0 [84.2 to 99.9]
  Additional serotype 5 | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 6A | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 7F | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 19A | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 4: difference in proportions, [(7vPnC/13vPnC) - (MnCC/13vPnC)], expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 6B: difference in proportions, [(7vPnC/13vPnC) - (MnCC/13vPnC)], expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 9V: difference in proportions, [(7vPnC/13vPnC) - (MnCC/13vPnC)], expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 14: difference in proportions, [(7vPnC/13vPnC) - (MnCC/13vPnC)], expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = 2.9, 95% CI 2-sided [-6.9 to 14.9]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 18C: difference in proportions, [(7vPnC/13vPnC) - (MnCC/13vPnC)], expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 19F: difference in proportions, [(7vPnC/13vPnC) - (MnCC/13vPnC)], expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.4 to 10.3]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 23F: difference in proportions, [(7vPnC/13vPnC) - (MnCC/13vPnC)], expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 1: difference in proportions, [(7vPnC/13vPnC) - (MnCC/13vPnC)], expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 3: difference in proportions, [(7vPnC/13vPnC) - (MnCC/13vPnC)], expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = -2.2, 95% CI 2-sided [-15.7 to 10.9]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 5: difference in proportions, [(7vPnC/13vPnC) - (MnCC/13vPnC)], expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 6A: difference in proportions, [(7vPnC/13vPnC) - (MnCC/13vPnC)], expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 7F: difference in proportions, [(7vPnC/13vPnC) - (MnCC/13vPnC)], expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 19A: difference in proportions, [(7vPnC/13vPnC) - (MnCC/13vPnC)], expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]

2. Primary Outcome: Percentage of Participants Achieving a Pneumococcal IgG Antibody Concentration ≥0.35 Mcg/mL for the 13 Serotypes for 7vPnC / 13vPnC in Comparison to MnCC / 13vPnC After Vaccination (Visit 4)
Description: Percentage of participants achieving predefined IgG antibody threshold ≥0.35 Mcg/mL for the 13 pneumococcal serotypes (7vPnC serotypes 4, 6B, 9V, 14, 18C, 19F, 23F and additional serotypes 1, 3, 5, 6A, 7F, and 19A) along with the exact, 2-sided 95% CIs based on the observed percentage of participants.
Time Frame: Day 7 (Visit 4)
Population: Evaluable Immunogenicity population; N=number of participants with a determinate IgG antibody concentration for the serotypes.
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Number analyzed (Participants) | 38 | 35
observed percentage of participants
  7vPnC serotype 4 | 94.7 [82.3 to 99.4] | 85.7 [69.7 to 95.2]
  7vPnC serotype 6B | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  7vPnC serotype 9V | 100.0 [90.7 to 100.0] | 97.1 [85.1 to 99.9]
  7vPnC serotype 14 | 100.0 [90.7 to 100.0] | 94.3 [80.8 to 99.3]
  7vPnC serotype 18C | 97.4 [86.2 to 99.9] | 94.3 [80.8 to 99.3]
  7vPnC serotype 19F | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  7vPnC serotype 23F | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 1 | 100.0 [90.7 to 100.0] | 97.1 [85.1 to 99.9]
  Additional serotype 3 | 94.7 [82.3 to 99.4] | 87.9 [71.8 to 96.6]
  Additional serotype 5 | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 6A | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 7F | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 19A | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; difference in proportions = 9.0, 95% CI 2-sided [-5.6 to 25.5]
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; difference in proportions = 2.9, 95% CI 2-sided [-6.9 to 14.9]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; difference in proportions = 5.7, 95% CI 2-sided [-4.2 to 19.2]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; difference in proportions = 3.1, 95% CI 2-sided [-9.3 to 17.0]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.4 to 10.3]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; difference in proportions = 2.9, 95% CI 2-sided [-6.9 to 14.9]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; difference in proportions = 6.9, 95% CI 2-sided [-7.4 to 23.4]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]

3. Primary Outcome: Percentage of Participants Achieving a Pneumococcal Opsonophagocytic Activity (OPA) Antibody Titer ≥LLOQ for the 13 Serotypes for 7vPnC / 13vPnC in Comparison to MnCC / 13vPnC After Vaccination (Visit 5)
Description: Percentage of participants achieving predefined OPA antibody titer ≥ serotype-specific lower limit of quantification (LLOQ) using modified microcolony assays for the 13 pneumococcal serotypes (7vPnC serotypes 4, 6B, 9V, 14, 18C, 19F, 23F and additional serotypes 1, 3, 5, 6A, 7F, and 19A) along with the exact, 2-sided 95% CIs based on the observed percentage of participants. LLOQ for each serotype: 1=1:8, 3=1:12, 4=1:21, 5=1:29, 6A=1:37, 6B=1:43, 7F=1:210, 9V=1:345, 14=1:35, 18C=1:31, 19A=1:18, 19F=1:48, 23F=1:13.
Time Frame: Day 28 (Visit 5)
Population: Evaluable Immunogenicity population; N=number of participants with a determinate OPA antibody titer to the serotypes.
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Number analyzed (Participants) | 38 | 35
observed percentage of participants
  7vPnC serotype 4 | 100.0 [90.3 to 100.0] | 100.0 [89.1 to 100.0]
  7vPnC serotype 6B | 100.0 [90.5 to 100.0] | 100.0 [90.0 to 100.0]
  7vPnC serotype 9V | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  7vPnC serotype 14 | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  7vPnC serotype 18C | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  7vPnC serotype 19F | 97.4 [86.2 to 99.9] | 100.0 [89.7 to 100.0]
  7vPnC serotype 23F | 100.0 [90.5 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 1 | 100.0 [90.7 to 100.0] | 97.1 [84.7 to 99.9]
  Additional serotype 3 | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 5 | 89.5 [75.2 to 97.1] | 88.6 [73.3 to 96.8]
  Additional serotype 6A | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  Additional serotype 7F | 100.0 [90.5 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 19A | 97.4 [86.2 to 99.9] | 100.0 [90.0 to 100.0]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 4: difference in proportions, [7vPnC / 13vPnC) - (MnCC / 13vPnC), expressed as a percentage, along with exact 2-sided confidence interval; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.2 to 10.9]
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.0 to 10.1]
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.4 to 10.3]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.4 to 10.3]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; difference in proportions = -2.6, 95% CI 2-sided [-13.9 to 8.0]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.0 to 10.1]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; difference in proportions = 2.9, 95% CI 2-sided [-6.7 to 15.3]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; difference in proportions = 0.9, 95% CI 2-sided [-15.0 to 17.6]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.4 to 10.3]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.0 to 10.1]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; difference in proportions = -2.6, 95% CI 2-sided [-13.9 to 7.6]

4. Primary Outcome: Percentage of Participants Achieving a Pneumococcal Opsonophagocytic Activity (OPA) Antibody Titer ≥LLOQ for the 13 Serotypes for 7vPnC / 13vPnC in Comparison to MnCC / 13vPnC After Vaccination (Visit 4)
Description: as for outcome 3
Time Frame: Day 7 (Visit 4)
Population: Evaluable Immunogenicity population; N=number of participants with a determinate OPA antibody titer to the serotypes.
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Number analyzed (Participants) | 38 | 35
observed percentage of participants
  7vPnC serotype 4 | 97.4 [86.2 to 99.9] | 100.0 [89.7 to 100.0]
  7vPnC serotype 6B | 100.0 [90.7 to 100.0] | 100.0 [89.4 to 100.0]
  7vPnC serotype 9V | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  7vPnC serotype 14 | 100.0 [90.5 to 100.0] | 100.0 [89.7 to 100.0]
  7vPnC serotype 18C | 100.0 [90.5 to 100.0] | 100.0 [90.0 to 100.0]
  7vPnC serotype 19F | 94.3 [80.8 to 99.3] | 97.1 [84.7 to 99.9]
  7vPnC serotype 23F | 97.3 [85.8 to 99.9] | 94.3 [80.8 to 99.3]
  Additional serotype 1 | 100.0 [90.5 to 100.0] | 97.1 [85.1 to 99.9]
  Additional serotype 3 | 97.4 [86.2 to 99.9] | 100.0 [89.7 to 100.0]
  Additional serotype 5 | 89.5 [75.2 to 97.1] | 88.2 [72.5 to 96.7]
  Additional serotype 6A | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 7F | 100.0 [90.5 to 100.0] | 97.0 [84.2 to 99.9]
  Additional serotype 19A | 97.4 [86.2 to 99.9] | 100.0 [90.0 to 100.0]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; difference in proportions = -2.6, 95% CI 2-sided [-13.9 to 8.0]
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.2 to 10.6]
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.4 to 10.3]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.3]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.0 to 10.1]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; difference in proportions = -2.8, 95% CI 2-sided [-16.8 to 10.1]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; difference in proportions = 3.0, 95% CI 2-sided [-9.1 to 16.6]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; difference in proportions = 2.9, 95% CI 2-sided [-7.1 to 15.0]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; difference in proportions = -2.6, 95% CI 2-sided [-13.9 to 8.0]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; difference in proportions = 1.2, 95% CI 2-sided [-14.8 to 18.2]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; difference in proportions = 3.0, 95% CI 2-sided [-6.8 to 15.8]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; difference in proportions = -2.6, 95% CI 2-sided [-13.9 to 7.6]

5. Secondary Outcome: Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for the 13 Serotypes Relative to 7vPnC / 13vPnC Prevaccination Visit 1 and Postvaccination Visit 5
Description: Pneumococcal IgG GMCs measured as Mcg/mL for the 13 pneumococcal serotypes (7vPnC serotypes 4, 6B, 9V, 14, 18C, 19F, 23F and additional serotypes 1, 3, 5, 6A, 7F, and 19A). The 2-sided, 95% CIs for the GMCs were constructed by back transformation of the CIs for the mean of the logarithmically transformed assay results computed using the Student t distribution.
Time Frame: Baseline (Visit 1), Day 28 (Visit 5)
Population: Evaluable Immunogenicity population. GMCs calculated using all participants with available data at both the prevaccination and postvaccination blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: Mcg/mL
Groups:
- 7vPnC / 13vPnC Prevaccination Visit 1; 7vPnC / 13vPnC Postvaccination Visit 5: 13vPnC administered as a single 0.5 mL dose IM. Participants had previously received 7vPnC in study D118-P8.
Arm/Group | 7vPnC / 13vPnC Prevaccination Visit 1 | 7vPnC / 13vPnC Postvaccination Visit 5
Number analyzed (Participants) | 38 | 38
Mcg/mL
  7vPnC serotype 4 | 0.20 [0.12 to 0.33] | 5.96 [4.10 to 8.65]
  7vPnC serotype 6B | 5.89 [4.61 to 7.51] | 66.72 [50.19 to 88.70]
  7vPnC serotype 9V | 1.54 [1.19 to 2.00] | 8.62 [6.55 to 11.34]
  7vPnC serotype 14 | 0.58 [0.39 to 0.86] | 41.45 [27.72 to 61.97]
  7vPnC serotype 18C | 0.75 [0.48 to 1.18] | 5.93 [4.34 to 8.11]
  7vPnC serotype 19F | 2.94 [2.08 to 4.15] | 13.41 [8.89 to 20.23]
  7vPnC serotype 23F | 2.51 [1.92 to 3.27] | 17.20 [12.44 to 23.77]
  Additional serotype 1 | 1.04 [0.71 to 1.54] | 11.59 [7.34 to 18.30]
  Additional serotype 3 | 1.30 [0.83 to 2.04] | 2.19 [1.60 to 2.99]
  Additional serotype 5 | 3.24 [2.45 to 4.27] | 6.80 [4.75 to 9.74]
  Additional serotype 6A | 3.78 [2.85 to 5.03] | 29.11 [19.04 to 44.50]
  Additional serotype 7F | 1.38 [0.93 to 2.05] | 9.92 [7.03 to 14.01]
  Additional serotype 19A | 7.05 [5.52 to 8.99] | 21.29 [14.90 to 30.43]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; 7vPnC serotype 4: Geometric mean fold rises (GMFRs) were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 29.47, 95% CI 2-sided [17.61 to 49.33] — Confidence intervals (CI) for the GMRFs are back transformations of confidence levels based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; 7vPnC serotype 6B: GMFRs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 11.34, 95% CI 2-sided [8.49 to 15.13] — CIs for the GMRFs are back transformations of confidence levels based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; 7vPnC serotype 9V: GMFRs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 5.58, 95% CI 2-sided [4.06 to 7.67] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; 7vPnC serotype 14: GMFRs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 71.09, 95% CI 2-sided [40.74 to 124.08] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; 7vPnC serotype 18C: GMFRs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 7.91, 95% CI 2-sided [4.92 to 12.73] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; 7vPnC serotype 19F: GMFRs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 4.56, 95% CI 2-sided [2.87 to 7.26] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; 7vPnC serotype 23F: GMFRs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 6.85, 95% CI 2-sided [4.51 to 10.42] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; Additional serotype 1: GMFRs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 11.10, 95% CI 2-sided [6.98 to 17.64] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; Additional serotype 3: GMFRs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 1.68, 95% CI 2-sided [1.37 to 2.07] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; Additional serotype 5: GMFRs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 2.10, 95% CI 2-sided [1.52 to 2.90] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; Additional serotype 6A: GMFRs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 7.70, 95% CI 2-sided [4.77 to 12.42] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; Additional serotype 7F: GMFRs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 7.20, 95% CI 2-sided [4.95 to 10.48] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; Additional serotype 19A: GMFRs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 3.02, 95% CI 2-sided [2.23 to 4.10] — [estimate comment as in outcome 5, analysis 2]

6. Secondary Outcome: Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for the 13 Serotypes Relative to MnCC / 13vPnC Prevaccination Visit 1 and Postvaccination Visit 5
Description: as for outcome 5
Time Frame: Baseline (Visit 1), Day 28 (Visit 5)
Population: Evaluable Immunogenicity population; GMCs calculated using all participants with available data at both the prevaccination and postvaccination blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: Mcg/mL
Groups:
- MnCC / 13vPnC Prevaccination Visit 1; MnCC / 13vPnC Postvaccination Visit 5: 13vPnC administered as a single 0.5 mL dose IM. Participants had previously received MnCC in study D118-P8.
Arm/Group | MnCC / 13vPnC Prevaccination Visit 1 | MnCC / 13vPnC Postvaccination Visit 5
Number analyzed (Participants) | 35 | 35
Mcg/mL
  7vPnC serotype 4 | 0.15 [0.07 to 0.29] | 2.86 [2.00 to 4.07]
  7vPnC serotype 6B | 3.97 [2.78 to 5.67] | 22.62 [14.56 to 35.16]
  7vPnC serotype 9V | 1.69 [1.20 to 2.38] | 4.70 [3.49 to 6.33]
  7vPnC serotype 14 | 0.79 [0.43 to 1.43] | 18.50 [10.10 to 33.90]
  7vPnC serotype 18C | 0.72 [0.46 to 1.13] | 9.79 [6.43 to 14.90]
  7vPnC serotype 19F | 2.01 [1.32 to 3.05] | 18.02 [11.56 to 28.08]
  7vPnC serotype 23F | 2.31 [1.70 to 3.14] | 20.80 [13.07 to 33.08]
  Additional serotype 1 | 0.70 [0.43 to 1.15] | 5.30 [3.40 to 8.26]
  Additional serotype 3 | 1.16 [0.73 to 1.86] | 1.81 [1.25 to 2.62]
  Additional serotype 5 | 3.83 [2.77 to 5.31] | 7.39 [4.98 to 10.96]
  Additional serotype 6A | 3.82 [2.79 to 5.23] | 17.05 [10.82 to 26.87]
  Additional serotype 7F | 1.12 [0.73 to 1.72] | 5.94 [4.08 to 8.65]
  Additional serotype 19A | 6.18 [4.57 to 8.35] | 20.17 [15.28 to 26.63]
Statistical Analysis 1: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; 7vPnC serotype 4: GMFRs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 19.68, 95% CI 2-sided [9.99 to 38.77] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; geometric mean fold rise = 5.70, 95% CI 2-sided [3.90 to 8.33] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; geometric mean fold rise = 2.78, 95% CI 2-sided [2.16 to 3.57] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 4: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 23.46, 95% CI 2-sided [13.17 to 41.79] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 5: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; geometric mean fold rise = 13.68, 95% CI 2-sided [8.94 to 20.92] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 6: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; geometric mean fold rise = 8.98, 95% CI 2-sided [6.21 to 12.97] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 7: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 9.00, 95% CI 2-sided [5.91 to 13.72] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 8: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 8]; Test type: Superiority or Other; geometric mean fold rise = 7.58, 95% CI 2-sided [5.36 to 10.72] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 9: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 9]; Test type: Superiority or Other; geometric mean fold rise = 1.56, 95% CI 2-sided [1.30 to 1.86] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 10: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 1.93, 95% CI 2-sided [1.43 to 2.60] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 11: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; geometric mean fold rise = 4.46, 95% CI 2-sided [3.09 to 6.45] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 12: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 12]; Test type: Superiority or Other; geometric mean fold rise = 5.32, 95% CI 2-sided [3.65 to 7.75] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 13: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 3.27, 95% CI 2-sided [2.49 to 4.28] — [estimate comment as in outcome 5, analysis 2]

7. Secondary Outcome: Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for the 13 Serotypes Relative to 7vPnC / 13vPnC Prevaccination Visit 1 and Postvaccination Visit 4
Description: as for outcome 5
Time Frame: Baseline (Visit 1), Day 7 (Visit 4)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Mcg/mL
Groups:
- 7vPnC / 13vPnC Postvaccination Visit 4: 13vPnC administered as a single 0.5 mL dose IM. Participants had previously received 7vPnC in study D118-P8.
Arm/Group | 7vPnC / 13vPnC Prevaccination Visit 1 | 7vPnC / 13vPnC Postvaccination Visit 4
Number analyzed (Participants) | 38 | 38
Mcg/mL
  7vPnC serotype 4 | 0.20 [0.12 to 0.33] | 3.21 [2.10 to 4.90]
  7vPnC serotype 6B | 5.89 [4.61 to 7.51] | 29.46 [20.74 to 41.86]
  7vPnC serotype 9V | 1.54 [1.19 to 2.00] | 5.96 [4.57 to 7.76]
  7vPnC serotype 14 | 0.58 [0.39 to 0.86] | 10.25 [6.85 to 15.33]
  7vPnC serotype 18C | 0.75 [0.48 to 1.18] | 3.17 [2.26 to 4.42]
  7vPnC serotype 19F | 2.94 [2.08 to 4.15] | 7.46 [5.43 to 10.25]
  7vPnC serotype 23F | 2.51 [1.92 to 3.27] | 10.56 [7.69 to 14.51]
  Additional serotype 1 | 1.04 [0.71 to 1.54] | 4.42 [2.93 to 6.67]
  Additional serotype 3 | 1.30 [0.83 to 2.04] | 2.12 [1.54 to 2.92]
  Additional serotype 5 | 3.24 [2.45 to 4.27] | 5.40 [4.08 to 7.15]
  Additional serotype 6A | 3.78 [2.85 to 5.03] | 13.60 [9.01 to 20.53]
  Additional serotype 7F | 1.38 [0.93 to 2.05] | 4.70 [3.26 to 6.78]
  Additional serotype 19A | 7.05 [5.52 to 8.99] | 13.40 [10.30 to 17.42]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; 7vPnC serotype 4: GMFRs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 15.86, 95% CI 2-sided [9.16 to 27.46] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; 7vPnC serotype 6B: GMFRs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 5.01, 95% CI 2-sided [3.50 to 7.16] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; 7vPnC serotype 9V: GMFRs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 3.86, 95% CI 2-sided [2.93 to 5.09] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; 7vPnC serotype 14: GMFRs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 17.57, 95% CI 2-sided [11.11 to 27.79] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; 7vPnC serotype 18C: GMFRs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 4.22, 95% CI 2-sided [2.86 to 6.23] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; 7vPnC serotype 19F: GMFRs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 2.54, 95% CI 2-sided [1.78 to 3.62] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; 7vPnC serotype 23F: GMFRs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 4.21, 95% CI 2-sided [2.86 to 6.19] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; Additional serotype 1: GMFRs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 4.23, 95% CI 2-sided [2.79 to 6.42] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; Additional serotype 3: GMFRs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 1.63, 95% CI 2-sided [1.30 to 2.05] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; Additional serotype 5: GMFRs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 1.67, 95% CI 2-sided [1.30 to 2.14] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; Additional serotype 6A: GMFRs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 3.60, 95% CI 2-sided [2.39 to 5.42] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; Additional serotype 7F: GMFRs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 3.41, 95% CI 2-sided [2.42 to 4.82] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; Additional serotype 19A: GMFRs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 1.90, 95% CI 2-sided [1.60 to 2.26] — [estimate comment as in outcome 5, analysis 2]

8. Secondary Outcome: Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for the 13 Serotypes Relative to MnCC / 13vPnC Prevaccination Visit 1 and Postvaccination Visit 4
Description: as for outcome 5
Time Frame: Baseline (Visit 1), Day 7 (Visit 4)
Population: Evaluable Immunogenicity population; GMCs calculated using all participants with available data at both the prevaccination and postvaccination blood draws. N=number of participants with valid and determinate assay results for both the prevaccination and postvaccination blood draw.
Measure: Geometric Mean (95% Confidence Interval); unit: Mcg/mL
Groups:
- MnCC / 13vPnC Postvaccination Visit 4: 13vPnC administered as a single 0.5 mL dose IM. Participants had previously received MnCC in study D118-P8.
Arm/Group | MnCC / 13vPnC Prevaccination Visit 1 | MnCC / 13vPnC Postvaccination Visit 4
Number analyzed (Participants) | 35 | 35
Mcg/mL
  7vPnC serotype 4 | 0.15 [0.07 to 0.29] | 1.21 [0.70 to 2.11]
  7vPnC serotype 6B | 3.97 [2.78 to 5.67] | 9.42 [6.23 to 14.24]
  7vPnC serotype 9V | 1.69 [1.20 to 2.38] | 3.41 [2.51 to 4.65]
  7vPnC serotype 14 | 0.79 [0.43 to 1.43] | 5.22 [2.76 to 9.86]
  7vPnC serotype 18C | 0.72 [0.46 to 1.13] | 3.53 [2.16 to 5.76]
  7vPnC serotype 19F | 2.01 [1.32 to 3.05] | 5.47 [3.51 to 8.54]
  7vPnC serotype 23F | 2.31 [1.70 to 3.14] | 6.51 [4.24 to 10.01]
  Additional serotype 1 | 0.70 [0.43 to 1.15] | 2.65 [1.75 to 4.00]
  Additional serotype 3 | 1.11 [0.67 to 1.82] | 1.46 [0.97 to 2.20]
  Additional serotype 5 | 3.83 [2.77 to 5.31] | 5.00 [3.49 to 7.15]
  Additional serotype 6A | 3.82 [2.79 to 5.23] | 7.79 [5.17 to 11.72]
  Additional serotype 7F | 1.12 [0.73 to 1.72] | 3.21 [2.25 to 4.59]
  Additional serotype 19A | 6.18 [4.57 to 8.35] | 12.03 [8.83 to 16.39]
Statistical Analysis 1: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; geometric mean fold rise = 8.36, 95% CI 2-sided [4.50 to 15.56] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; geometric mean fold rise = 2.37, 95% CI 2-sided [1.78 to 3.16] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 3]; Test type: Superiority or Other; geometric mean fold rise = 2.02, 95% CI 2-sided [1.63 to 2.49] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 4: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 6.61, 95% CI 2-sided [4.31 to 10.15] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 5: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; geometric mean fold rise = 4.92, 95% CI 2-sided [3.34 to 7.26] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 6: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 6]; Test type: Superiority or Other; geometric mean fold rise = 2.73, 95% CI 2-sided [2.08 to 3.57] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 7: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 2.82, 95% CI 2-sided [2.08 to 3.83] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 8: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 8]; Test type: Superiority or Other; geometric mean fold rise = 3.79, 95% CI 2-sided [2.80 to 5.13] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 9: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 9]; Test type: Superiority or Other; geometric mean fold rise = 1.32, 95% CI 2-sided [1.11 to 1.57] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 10: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 1.30, 95% CI 2-sided [1.05 to 1.61] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 11: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 11]; Test type: Superiority or Other; geometric mean fold rise = 2.04, 95% CI 2-sided [1.51 to 2.75] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 12: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 12]; Test type: Superiority or Other; geometric mean fold rise = 2.87, 95% CI 2-sided [2.19 to 3.77] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 13: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 1.95, 95% CI 2-sided [1.59 to 2.39] — [estimate comment as in outcome 5, analysis 2]

9. Secondary Outcome: Pneumococcal Opsonophagocytic Activity (OPA) Assay Geometric Mean Titers (GMTs) for the 13 Serotypes Relative to 7vPnC / 13vPnC Prevaccination Visit 1 and Postvaccination Visit 5
Description: Antibody geometric mean titers as measured by opsonophagocytic activity (OPA) assay for 13 pneumococcal serotypes (7vPnC serotypes 4, 6B, 9V, 14, 18C, 19F, 23F and additional serotypes 1, 3, 5, 6A, 7F, and 19A). The 2-sided, 95% CIs for the GMTs were constructed by back transformation of the CIs for the mean of the logarithmically transformed assay results computed using the Student t distribution.
Time Frame: Baseline (Visit 1), Day 28 (Visit 5)
Population: Evaluable Immunogenicity population; GMTs calculated using all participants with available data at both the prevaccination and postvaccination blood draws.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 7vPnC / 13vPnC Prevaccination Visit 1 | 7vPnC / 13vPnC Postvaccination Visit 5
Number analyzed (Participants) | 38 | 38
Titer
  7vPnC serotype 4 | 22 [6.3 to 80.7] | 4535 [2836.5 to 7251.3]
  7vPnC serotype 6B | 1024 [488.4 to 2148.4] | 11939 [8748.1 to 16293.9]
  7vPnC serotype 9V | 43 [13.4 to 137.3] | 6709 [5097.5 to 8829.4]
  7vPnC serotype 14 | 159 [63.7 to 396.0] | 5946 [4361.1 to 8107.6]
  7vPnC serotype 18C | 54 [19.5 to 149.5] | 5067 [3375.1 to 7607.2]
  7vPnC serotype 19F | 33 [15.1 to 73.3] | 1623 [995.2 to 2647.9]
  7vPnC serotype 23F | 87 [34.1 to 223.4] | 2799 [2048.5 to 3823.2]
  Additional serotype 1 | 6 [4.3 to 7.4] | 440 [301.8 to 641.2]
  Additional serotype 3 | 11 [6.9 to 16.6] | 111 [87.1 to 141.1]
  Additional serotype 5 | 4 [3.6 to 5.6] | 277 [145.2 to 526.4]
  Additional serotype 6A | 17 [7.1 to 39.7] | 9029 [6255.0 to 13034.0]
  Additional serotype 7F | 60 [17.7 to 205.3] | 7036 [4886.0 to 10131.8]
  Additional serotype 19A | 76 [36.7 to 157.5] | 1869 [1099.8 to 3177.3]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; geometric mean fold rise = 201.8, 95% CI 2-sided [55.11 to 739.05] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; geometric mean fold rise = 11.7, 95% CI 2-sided [5.20 to 26.10] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; geometric mean fold rise = 156.4, 95% CI 2-sided [48.72 to 501.86] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 37.4, 95% CI 2-sided [13.71 to 102.31] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; geometric mean fold rise = 93.9, 95% CI 2-sided [30.99 to 284.31] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; geometric mean fold rise = 48.7, 95% CI 2-sided [23.27 to 101.97] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 32.1, 95% CI 2-sided [11.99 to 85.81] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 8]; Test type: Superiority or Other; geometric mean fold rise = 78.1, 95% CI 2-sided [50.42 to 120.94] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 9]; Test type: Superiority or Other; geometric mean fold rise = 10.3, 95% CI 2-sided [6.80 to 15.72] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 61.7, 95% CI 2-sided [32.75 to 116.34] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; geometric mean fold rise = 536.5, 95% CI 2-sided [212.04 to 1357.19] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 12]; Test type: Superiority or Other; geometric mean fold rise = 116.9, 95% CI 2-sided [33.28 to 410.33] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 24.6, 95% CI 2-sided [11.30 to 53.42] — [estimate comment as in outcome 5, analysis 2]

10. Secondary Outcome: Pneumococcal Opsonophagocytic Activity (OPA) Assay Geometric Mean Titers (GMTs) for the 13 Serotypes Relative to MnCC / 13vPnC Prevaccination Visit 1 and Postvaccination Visit 5
Description: as for outcome 9
Time Frame: Baseline (Visit 1), Day 28 (Visit 5)
Population: Evaluable Immunogenicity population; GMTs calculated using all participants with available data at both the prevaccination and postvaccination blood draws. N=number of participants with valid and determinate assay results for both the prevaccination and postvaccination blood draw.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MnCC / 13vPnC Prevaccination Visit 1 | MnCC / 13vPnC Postvaccination Visit 5
Number analyzed (Participants) | 35 | 35
Titer
  7vPnC serotype 4 | 28 [4.5 to 174.3] | 4704 [2958.0 to 7481.1]
  7vPnC serotype 6B | 288 [74.8 to 1106.9] | 11607 [7762.6 to 17354.1]
  7vPnC serotype 9V | 120 [37.9 to 382.8] | 7457 [5702.3 to 9751.9]
  7vPnC serotype 14 | 262 [98.1 to 700.5] | 7006 [4997.7 to 9822.1]
  7vPnC serotype 18C | 25 [8.4 to 75.7] | 5736 [4141.4 to 7943.8]
  7vPnC serotype 19F | 23 [10.5 to 50.6] | 2696 [1831.0 to 3968.5]
  7vPnC serotype 23F | 11 [5.0 to 23.5] | 5197 [3599.2 to 7503.1]
  Additional serotype 1 | 5 [4.0 to 6.6] | 341 [221.9 to 524.9]
  Additional serotype 3 | 11 [7.0 to 18.2] | 98 [75.2 to 126.9]
  Additional serotype 5 | 4 [3.7 to 5.0] | 336 [175.4 to 642.2]
  Additional serotype 6A | 24 [8.9 to 64.2] | 10488 [7460.6 to 14744.7]
  Additional serotype 7F | 76 [21.1 to 275.2] | 6098 [4392.9 to 8464.9]
  Additional serotype 19A | 39 [19.9 to 78.1] | 2424 [1696.6 to 3462.4]
Statistical Analysis 1: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; geometric mean fold rise = 168.8, 95% CI 2-sided [20.22 to 1409.76] — CI for the GMRFs are back transformations of confidence levels based on the Student t distribution for the mean logarithm of the mean fold rise
Statistical Analysis 2: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; 7vPnC serotype 6B: GMRFs were calculated (postvaccination Visit 5 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 40.3, 95% CI 2-sided [10.97 to 148.44] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; geometric mean fold rise = 61.9, 95% CI 2-sided [18.83 to 203.72] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 4: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 26.7, 95% CI 2-sided [9.67 to 73.84] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 5: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; geometric mean fold rise = 226.9, 95% CI 2-sided [79.81 to 645.29] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 6: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; geometric mean fold rise = 116.8, 95% CI 2-sided [54.54 to 250.13] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 7: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 481.0, 95% CI 2-sided [207.01 to 1117.69] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 8: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 8]; Test type: Superiority or Other; geometric mean fold rise = 66.5, 95% CI 2-sided [41.80 to 105.75] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 9: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 9]; Test type: Superiority or Other; geometric mean fold rise = 8.6, 95% CI 2-sided [5.36 to 13.94] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 10: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 78.2, 95% CI 2-sided [41.38 to 147.80] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 11: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 11]; Test type: Superiority or Other; geometric mean fold rise = 438.1, 95% CI 2-sided [169.52 to 1132.43] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 12: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 12]; Test type: Superiority or Other; geometric mean fold rise = 80.0, 95% CI 2-sided [23.28 to 274.82] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 13: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 5; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 61.5, 95% CI 2-sided [28.73 to 131.76] — [estimate comment as in outcome 5, analysis 2]

11. Secondary Outcome: Pneumococcal Opsonophagocytic Activity (OPA) Assay Geometric Mean Titers (GMTs) for the 13 Serotypes Relative to 7vPnC / 13vPnC Prevaccination Visit 1 and Postvaccination Visit 4
Description: as for outcome 9
Time Frame: Baseline (Visit 1), Day 7 (Visit 4)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 7vPnC / 13vPnC Prevaccination Visit 1 | 7vPnC / 13vPnC Postvaccination Visit 4
Number analyzed (Participants) | 37 | 37
Titer
  7vPnC serotype 4 | 19 [6.0 to 62.8] | 5449 [3118.6 to 9519.8]
  7vPnC serotype 6B | 1034 [505.1 to 2116.9] | 7885 [5792.0 to 10734.0]
  7vPnC serotype 9V | 43 [13.4 to 137.3] | 6497 [4357.4 to 9687.5]
  7vPnC serotype 14 | 148 [58.2 to 375.7] | 3497 [2440.8 to 5009.1]
  7vPnC serotype 18C | 58 [20.6 to 163.8] | 5922 [3784.0 to 9268.9]
  7vPnC serotype 19F | 40 [17.4 to 91.6] | 1243 [620.6 to 2489.8]
  7vPnC serotype 23F | 79 [31.4 to 201.3] | 1487 [884.7 to 2499.5]
  Additional serotype 1 | 6 [4.3 to 7.6] | 367 [228.8 to 587.3]
  Additional serotype 3 | 11 [6.9 to 16.6] | 119 [82.1 to 172.0]
  Additional serotype 5 | 4 [3.6 to 5.6] | 185 [100.9 to 337.5]
  Additional serotype 6A | 17 [7.1 to 39.7] | 8072 [5195.8 to 12538.8]
  Additional serotype 7F | 60 [17.7 to 205.3] | 4601 [2998.3 to 7060.6]
  Additional serotype 19A | 76 [36.7 to 157.5] | 1345 [767.4 to 2357.7]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; geometric mean fold rise = 281.7, 95% CI 2-sided [76.65 to 1035.49] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 2]; Test type: Superiority or Other; geometric mean fold rise = 7.6, 95% CI 2-sided [3.47 to 16.75] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 3]; Test type: Superiority or Other; geometric mean fold rise = 151.4, 95% CI 2-sided [42.01 to 545.84] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 23.7, 95% CI 2-sided [8.67 to 64.54] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; geometric mean fold rise = 102.1, 95% CI 2-sided [32.00 to 325.40] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 6]; Test type: Superiority or Other; geometric mean fold rise = 31.1, 95% CI 2-sided [12.71 to 76.13] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 18.7, 95% CI 2-sided [6.82 to 51.39] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 8]; Test type: Superiority or Other; geometric mean fold rise = 64.4, 95% CI 2-sided [37.33 to 111.18] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 9]; Test type: Superiority or Other; geometric mean fold rise = 11.1, 95% CI 2-sided [6.64 to 18.52] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 41.2, 95% CI 2-sided [23.09 to 73.48] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 11]; Test type: Superiority or Other; geometric mean fold rise = 479.6, 95% CI 2-sided [171.63 to 1339.96] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 12]; Test type: Superiority or Other; geometric mean fold rise = 76.4, 95% CI 2-sided [21.63 to 270.02] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC Prevaccination Visit 1 vs 7vPnC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 17.7, 95% CI 2-sided [7.61 to 41.08] — [estimate comment as in outcome 5, analysis 2]

12. Secondary Outcome: Pneumococcal Opsonophagocytic Activity (OPA) Assay Geometric Mean Titers (GMTs) for the 13 Serotypes Relative to MnCC / 13vPnC Prevaccination Visit 1 and Postvaccination Visit 4
Description: as for outcome 9
Time Frame: Baseline (Visit 1), Day 7 (Visit 4)
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | MnCC / 13vPnC Prevaccination Visit 1 | MnCC / 13vPnC Postvaccination Visit 4
Number analyzed (Participants) | 34 | 34
Titer
  7vPnC serotype 4 | 40 [6.3 to 254.0] | 6782 [3687.6 to 12471.3]
  7vPnC serotype 6B | 405 [103.5 to 1584.7] | 7195 [4585.5 to 11289.8]
  7vPnC serotype 9V | 116 [36.8 to 364.9] | 7855 [5532.9 to 11152.1]
  7vPnC serotype 14 | 280 [103.1 to 760.7] | 6209 [4253.9 to 9063.3]
  7vPnC serotype 18C | 25 [8.4 to 75.7] | 5193 [3658.1 to 7372.3]
  7vPnC serotype 19F | 20 [9.4 to 44.7] | 1855 [1055.8 to 3258.2]
  7vPnC serotype 23F | 11 [5.0 to 23.5] | 991 [501.3 to 1959.3]
  Additional serotype 1 | 5 [4.0 to 6.5] | 385 [249.4 to 595.6]
  Additional serotype 3 | 12 [7.2 to 19.0] | 101 [72.2 to 141.7]
  Additional serotype 5 | 4 [3.7 to 5.0] | 258 [132.3 to 503.4]
  Additional serotype 6A | 23 [8.7 to 59.1] | 6107 [4149.7 to 8987.5]
  Additional serotype 7F | 95 [24.7 to 363.8] | 3577 [1774.8 to 7208.2]
  Additional serotype 19A | 39 [19.9 to 78.1] | 1763 [1220.1 to 2547.6]
Statistical Analysis 1: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; geometric mean fold rise = 170.2, 95% CI 2-sided [22.24 to 1301.79] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; 7vPnC serotype 6B: GMRFs were calculated (postvaccination Visit 4 / prevaccination Visit 1) using all participants with available data from both the prevaccination and postvaccination blood draws; Test type: Superiority or Other; geometric mean fold rise = 17.8, 95% CI 2-sided [5.27 to 59.91] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 3]; Test type: Superiority or Other; geometric mean fold rise = 67.8, 95% CI 2-sided [18.45 to 249.02] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 4: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 4]; Test type: Superiority or Other; geometric mean fold rise = 22.2, 95% CI 2-sided [7.94 to 61.88] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 5: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 5]; Test type: Superiority or Other; geometric mean fold rise = 205.5, 95% CI 2-sided [70.04 to 602.78] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 6: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 6]; Test type: Superiority or Other; geometric mean fold rise = 90.5, 95% CI 2-sided [40.28 to 203.27] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 7: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 7]; Test type: Superiority or Other; geometric mean fold rise = 91.7, 95% CI 2-sided [36.25 to 232.13] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 8: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 8]; Test type: Superiority or Other; geometric mean fold rise = 75.6, 95% CI 2-sided [47.32 to 120.91] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 9: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 9]; Test type: Superiority or Other; geometric mean fold rise = 8.7, 95% CI 2-sided [5.21 to 14.40] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 10: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 10]; Test type: Superiority or Other; geometric mean fold rise = 60.0, 95% CI 2-sided [31.06 to 115.92] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 11: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 11]; Test type: Superiority or Other; geometric mean fold rise = 269.8, 95% CI 2-sided [105.09 to 692.60] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 12: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 12]; Test type: Superiority or Other; geometric mean fold rise = 37.7, 95% CI 2-sided [10.85 to 131.09] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 13: Comparison: MnCC / 13vPnC Prevaccination Visit 1 vs MnCC / 13vPnC Postvaccination Visit 4; [analysis description as in outcome 7, analysis 13]; Test type: Superiority or Other; geometric mean fold rise = 44.8, 95% CI 2-sided [21.31 to 94.01] — [estimate comment as in outcome 5, analysis 2]

13. Secondary Outcome: Comparison of Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for the 13 Serotypes for 7vPnC / 13vPnC Relative to MnCC / 13vPnC After Vaccination (Visit 5)
Description: as for outcome 5
Time Frame: Day 28 (Visit 5)
Population: Evaluable Immunogenicity population; GMCs were calculated using all participants with available data for the specified blood draw. N=number of participants with a determinate OPA antibody concentration for the serotypes.
Measure: Geometric Mean (95% Confidence Interval); unit: Mcg/mL
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Number analyzed (Participants) | 38 | 35
Mcg/mL
  7vPnC serotype 4 | 5.73 [4.21 to 7.81] | 2.92 [2.22 to 3.83]
  7vPnC serotype 6B | 66.72 [50.19 to 88.70] | 22.62 [14.56 to 35.16]
  7vPnC serotype 9V | 8.72 [6.68 to 11.40] | 4.70 [3.49 to 6.33]
  7vPnC serotype 14 | 41.45 [27.72 to 61.97] | 18.50 [10.10 to 33.90]
  7vPnC serotype 18C | 5.72 [4.18 to 7.82] | 9.04 [5.98 to 13.68]
  7vPnC serotype 19F | 14.17 [9.54 to 21.07] | 15.80 [10.00 to 24.96]
  7vPnC serotype 23F | 17.20 [12.44 to 23.77] | 20.80 [13.07 to 33.08]
  Additional serotype 1 | 9.55 [6.46 to 14.13] | 5.63 [3.67 to 8.64]
  Additional serotype 3 | 2.13 [1.58 to 2.87] | 1.71 [1.20 to 2.44]
  Additional serotype 5 | 6.80 [4.75 to 9.74] | 7.52 [5.12 to 11.04]
  Additional serotype 6A | 29.11 [19.04 to 44.50] | 16.08 [10.18 to 25.40]
  Additional serotype 7F | 9.92 [7.03 to 14.01] | 5.75 [3.98 to 8.33]
  Additional serotype 19A | 21.29 [14.90 to 30.43] | 20.17 [15.28 to 26.63]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 4: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.97, 95% CI 2-sided [1.31 to 2.95] — CIs for the ratio are back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures [(7vPnC/13vPnC) - (MnCC/13vPnC)]
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 6B: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 2.95, 95% CI 2-sided [1.78 to 4.90] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 9V: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.85, 95% CI 2-sided [1.25 to 2.75] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 14: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 2.24, 95% CI 2-sided [1.11 to 4.53] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 18C: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 0.63, 95% CI 2-sided [0.38 to 1.05] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 19F: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 0.90, 95% CI 2-sided [0.50 to 1.62] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 23F: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 0.83, 95% CI 2-sided [0.48 to 1.43] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 1: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.70, 95% CI 2-sided [0.96 to 3.00] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 3: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.25, 95% CI 2-sided [0.79 to 1.96] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 5: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 0.90, 95% CI 2-sided [0.54 to 1.52] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 6A: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.81, 95% CI 2-sided [0.98 to 3.34] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 7F: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.72, 95% CI 2-sided [1.05 to 2.83] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 19A: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.06, 95% CI 2-sided [0.67 to 1.66] — [estimate comment as in outcome 13, analysis 1]

14. Secondary Outcome: Comparison of Pneumococcal Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for the 13 Serotypes for 7vPnC / 13vPnC Relative to MnCC / 13vPnC After Vaccination (Visit 4)
Description: as for outcome 5
Time Frame: Day 7 (Visit 4)
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Mcg/mL
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Number analyzed (Participants) | 38 | 35
Mcg/mL
  7vPnC serotype 4 | 3.00 [2.07 to 4.35] | 1.37 [0.90 to 2.10]
  7vPnC serotype 6B | 29.46 [20.74 to 41.86] | 9.42 [6.23 to 14.24]
  7vPnC serotype 9V | 5.75 [4.40 to 7.51] | 3.41 [2.51 to 4.65]
  7vPnC serotype 14 | 10.25 [6.85 to 15.33] | 5.22 [2.76 to 9.86]
  7vPnC serotype 18C | 3.09 [2.22 to 4.29] | 3.45 [2.16 to 5.52]
  7vPnC serotype 19F | 7.66 [5.66 to 10.36] | 4.85 [3.09 to 7.62]
  7vPnC serotype 23F | 10.56 [7.69 to 14.51] | 6.51 [4.24 to 10.01]
  Additional serotype 1 | 3.98 [2.82 to 5.62] | 2.83 [1.86 to 4.32]
  Additional serotype 3 | 2.02 [1.48 to 2.76] | 1.40 [0.95 to 2.06]
  Additional serotype 5 | 5.40 [4.08 to 7.15] | 5.12 [3.60 to 7.28]
  Additional serotype 6A | 13.60 [9.01 to 20.53] | 7.25 [4.75 to 11.06]
  Additional serotype 7F | 4.70 [3.26 to 6.78] | 3.17 [2.24 to 4.48]
  Additional serotype 19A | 13.40 [10.30 to 17.42] | 12.03 [8.83 to 16.39]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 4: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 2.18, 95% CI 2-sided [1.26 to 3.79] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 6B: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 3.13, 95% CI 2-sided [1.84 to 5.32] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 9V: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.68, 95% CI 2-sided [1.13 to 2.51] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 14: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.96, 95% CI 2-sided [0.95 to 4.07] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 18C: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 0.90, 95% CI 2-sided [0.51 to 1.56] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 19F: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.58, 95% CI 2-sided [0.93 to 2.66] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 23F: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.62, 95% CI 2-sided [0.97 to 2.73] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 1: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.41, 95% CI 2-sided [0.83 to 2.39] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 3: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.44, 95% CI 2-sided [0.89 to 2.34] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 5: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.06, 95% CI 2-sided [0.68 to 1.64] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 6A: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.88, 95% CI 2-sided [1.05 to 3.35] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 7F: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.48, 95% CI 2-sided [0.90 to 2.44] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 19A: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean concentrations = 1.11, 95% CI 2-sided [0.75 to 1.66] — [estimate comment as in outcome 13, analysis 1]

15. Secondary Outcome: Comparison of Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for the 13 Serotypes for 7vPnC / 13vPnC Relative to MnCC / 13vPnC After Vaccination (Visit 5)
Description: as for outcome 9
Time Frame: Day 28 (Visit 5)
Population: Evaluable Immunogenicity population; GMTs were calculated using all participants with available data for the specified blood draw. N=number of participants with a determinate OPA antibody titer for the serotypes.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Number analyzed (Participants) | 38 | 35
Titer
  7vPnC serotype 4 | 4626 [3322.5 to 6441.2] | 6065 [4590.9 to 8012.5]
  7vPnC serotype 6B | 11451 [8290.4 to 15817.9] | 10380 [7515.2 to 14336.9]
  7vPnC serotype 9V | 6346 [5152.2 to 7817.5] | 7555 [5916.7 to 9646.8]
  7vPnC serotype 14 | 5898 [4481.0 to 7762.1] | 7031 [5195.6 to 9515.5]
  7vPnC serotype 18C | 5090 [3428.4 to 7557.7] | 6005 [4389.3 to 8214.6]
  7vPnC serotype 19F | 1623 [995.2 to 2647.9] | 2696 [1831.0 to 3968.5]
  7vPnC serotype 23F | 2752 [2074.6 to 3651.3] | 4841 [3574.5 to 6555.1]
  Additional serotype 1 | 449 [312.8 to 643.2] | 347 [228.3 to 527.4]
  Additional serotype 3 | 113 [89.2 to 143.5] | 99 [77.0 to 126.3]
  Additional serotype 5 | 296 [158.8 to 549.9] | 336 [175.4 to 642.2]
  Additional serotype 6A | 9458 [6674.2 to 13404.0] | 10842 [7904.9 to 14870.9]
  Additional serotype 7F | 6740 [4933.2 to 9207.7] | 6050 [4515.0 to 8106.7]
  Additional serotype 19A | 2120 [1308.0 to 3435.3] | 2340 [1667.0 to 3285.4]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 4: ratio of GMTs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.8, 95% CI 2-sided [0.50 to 1.17] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 6B: ratio of GMTs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 1.1, 95% CI 2-sided [0.70 to 1.73] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 9V: ratio of GMTs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.8, 95% CI 2-sided [0.61 to 1.15] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 14: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.8, 95% CI 2-sided [0.56 to 1.25] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 18C: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.8, 95% CI 2-sided [0.51 to 1.40] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 19F: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.6, 95% CI 2-sided [0.32 to 1.12] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 23F: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.6, 95% CI 2-sided [0.38 to 0.85] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 1: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 1.3, 95% CI 2-sided [0.75 to 2.22] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 3: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 1.1, 95% CI 2-sided [0.82 to 1.61] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 5: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.9, 95% CI 2-sided [0.36 to 2.13] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 6A: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.9, 95% CI 2-sided [0.55 to 1.39] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 7F: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 1.1, 95% CI 2-sided [0.73 to 1.70] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 19A: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.9, 95% CI 2-sided [0.50 to 1.63] — [estimate comment as in outcome 13, analysis 1]

16. Secondary Outcome: Comparison of Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for the 13 Serotypes for 7vPnC / 13vPnC Relative to MnCC / 13vPnC After Vaccination (Visit 4)
Description: as for outcome 9
Time Frame: Day 7 (Visit 4)
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Number analyzed (Participants) | 38 | 35
Titer
  7vPnC serotype 4 | 5567 [3202.5 to 9678.7] | 8339 [6154.1 to 11299.5]
  7vPnC serotype 6B | 8082 [5743.5 to 11372.6] | 6450 [4477.8 to 9290.2]
  7vPnC serotype 9V | 6865 [4826.7 to 9763.7] | 7806 [5491.4 to 11095.6]
  7vPnC serotype 14 | 3596 [2613.0 to 4948.5] | 5994 [4246.9 to 8460.1]
  7vPnC serotype 18C | 5833 [3770.5 to 9023.7] | 5266 [3779.3 to 7338.4]
  7vPnC serotype 19F | 1243 [620.6 to 2489.8] | 1855 [1055.8 to 3258.2]
  7vPnC serotype 23F | 1575 [987.7 to 2511.7] | 1141 [655.1 to 1986.8]
  Additional serotype 1 | 379 [241.8 to 594.9] | 393 [257.2 to 600.3]
  Additional serotype 3 | 117 [81.3 to 167.5] | 104 [75.4 to 143.4]
  Additional serotype 5 | 200 [111.2 to 358.6] | 258 [132.3 to 503.4]
  Additional serotype 6A | 8534 [5631.9 to 12931.6] | 6199 [4357.6 to 8818.6]
  Additional serotype 7F | 4750 [3291.8 to 6852.9] | 3760 [2106.7 to 6709.5]
  Additional serotype 19A | 1504 [911.2 to 2484.1] | 1761 [1242.8 to 2496.0]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 4: ratio of GMTs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.7, 95% CI 2-sided [0.35 to 1.27] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 6B: ratio of GMTs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 1.3, 95% CI 2-sided [0.77 to 2.05] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 9V: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.9, 95% CI 2-sided [0.54 to 1.44] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 14: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.6, 95% CI 2-sided [0.38 to 0.95] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 18C: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 1.1, 95% CI 2-sided [0.64 to 1.91] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 19F: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.7, 95% CI 2-sided [0.28 to 1.62] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; 7vPnC serotype 23F: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 1.4, 95% CI 2-sided [0.68 to 2.81] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 1: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 1.0, 95% CI 2-sided [0.53 to 1.77] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 3: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 1.1, 95% CI 2-sided [0.69 to 1.81] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 5: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.8, 95% CI 2-sided [0.32 to 1.85] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 6A: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 1.4, 95% CI 2-sided [0.80 to 2.36] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 7F: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 1.3, 95% CI 2-sided [0.65 to 2.44] — [estimate comment as in outcome 13, analysis 1]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; Additional serotype 19A: ratio of GMCs for (7vPnC/13vPnC) relative to (MnCC/13vPnC); Test type: Superiority or Other; ratio of geometric mean titers = 0.9, 95% CI 2-sided [0.46 to 1.57] — [estimate comment as in outcome 13, analysis 1]

17. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Local Reactions Within 4 Days After Vaccination
Description: Local reactions reported using the diary card during the 4-day reactogenicity period after vaccination. Tenderness at injection site scaled as Any (tenderness present) or Significant (present and interfered with limb movement). Redness and swelling at injection site scaled as Any (redness or swelling present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); or Severe (> 7.0 cm). Participants may be represented in >1 category.
Time Frame: Baseline up to 4 days after vaccination on Day 1
Population: Safety population included all participants who received the vaccine. N=number of participants with analyzable data for reactogenicity events (reported Yes for at least 1 day or No for all days).
Measure: Number; unit: percentage of participants
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Number analyzed (Participants) | 38 | 36
percentage of participants
  Tenderness: Any | 92.1 | 86.1
  Tenderness: Significant | 10.5 | 19.4
  Swelling: Any | 10.5 | 5.6
  Swelling: Mild | 2.6 | 2.8
  Swelling: Moderate | 10.5 | 2.8
  Redness: Any | 5.3 | 5.6
  Redness: Mild | 0.0 | 2.8
  Redness: Moderate | 5.3 | 2.8

18. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-specified Systemic Events Within 4 Days After Vaccination
Description: Systemic events reported using the diary card during the 4-day reactogenicity period after vaccination. Temperature scaled as Fever ≥38 but ≤39 degrees Celsius (C) (mild), >39 but ≤40 degrees C (moderate), or >40 degrees C (severe). Presence of Decreased appetite, Irritability, Increased sleep, Decreased sleep, Rash, and Hives; also scaled as Mild (easily tolerated, minimal discomfort; not interfering with activities), Moderate (sufficiently discomforting to interfere with normal activities), or Severe (may prevent normal activities and require medical intervention).
Time Frame: Baseline up to 4 days after vaccination on Day 1
Population: Safety population; N=number of participants with analyzable data for reactogenicity events (reported Yes for at least 1 day or No for all days).
Measure: Number; unit: percentage of participants
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Number analyzed (Participants) | 38 | 36
percentage of participants
  Fever ≥38 but ≤39 degrees C | 2.9 | 0.0
  Decreased appetite | 7.9 | 16.7
  Decreased appetite: Mild | 7.9 | 11.1
  Decreased appetite: Moderate | 2.6 | 8.3
  Irritability | 18.4 | 13.9
  Irritability: Mild | 13.2 | 11.1
  Irritability: Moderate | 5.3 | 5.6
  Increased sleep | 26.3 | 33.3
  Increased sleep: Mild | 15.8 | 25.0
  Increased sleep: Moderate | 13.2 | 13.9
  Increased sleep: Severe | 2.6 | 0.0
  Decreased sleep | 7.9 | 11.1
  Decreased sleep: Mild | 5.3 | 8.3
  Decreased sleep: Moderate | 2.6 | 2.8
  Rash | 5.3 | 0.0
  Rash: Mild | 5.3 | 0.0

19. Primary Outcome: Percentage of Participants Achieving a Pneumococcal Opsonophagocytic Activity (OPA) Antibody Titer ≥1:8 for the 13 Serotypes for 7vPnC / 13vPnC in Comparison to MnCC / 13vPnC After Vaccination (Visit 5)
Description: Percentage of participants achieving predefined OPA antibody titer ≥1:8 for the 13 pneumococcal serotypes (7vPnC serotypes 4, 6B, 9V, 14, 18C, 19F, 23F and additional serotypes 1, 3, 5, 6A, 7F, and 19A) along with the exact, 2-sided 95% CIs based on the observed percentage of participants. The lowest titer that can be determined using the standard OPA assay is a titer of 1:8 limit of detection (LOD) and is the same for each serotype-specific OPA assay.
Time Frame: Day 28 (Visit 5)
Population: Evaluable Immunogenicity population; N=number of participants with a determinate OPA antibody titer to the serotypes.
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Number analyzed (Participants) | 38 | 35
observed percentage of participants
  7vPnC serotype 4 | 100.0 [90.3 to 100.0] | 100.0 [89.1 to 100.0]
  7vPnC serotype 6B | 100.0 [90.5 to 100.0] | 100.0 [90.0 to 100.0]
  7vPnC serotype 9V | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  7vPnC serotype 14 | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  7vPnC serotype 18C | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  7vPnC serotype 19F | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  7vPnC serotype 23F | 100.0 [90.5 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 1 | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  Additional serotype 3 | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 5 | 97.4 [86.2 to 99.9] | 94.3 [80.8 to 99.3]
  Additional serotype 6A | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  Additional serotype 7F | 100.0 [90.5 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 19A | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.2 to 10.9]
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.0 to 10.1]
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.4 to 10.3]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.4 to 10.3]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.4 to 10.3]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.0 to 10.1]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.4 to 10.3]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; difference in proportions = 3.1, 95% CI 2-sided [-9.3 to 17.0]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.4 to 10.3]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.0 to 10.1]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]

20. Primary Outcome: Percentage of Participants Achieving a Pneumococcal Opsonophagocytic Activity (OPA) Antibody Titer ≥1:8 for the 13 Serotypes for 7vPnC / 13vPnC in Comparison to MnCC / 13vPnC After Vaccination (Visit 4)
Description: as for outcome 19
Time Frame: Day 7 (Visit 4)
Population: Evaluable Immunogenicity population; N=number of participants with a determinate OPA antibody titer to the serotypes.
Measure: Number (95% Confidence Interval); unit: observed percentage of participants
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Number analyzed (Participants) | 38 | 35
observed percentage of participants
  7vPnC serotype 4 | 97.4 [86.2 to 99.9] | 100.0 [89.7 to 100.0]
  7vPnC serotype 6B | 100.0 [90.7 to 100.0] | 100.0 [89.4 to 100.0]
  7vPnC serotype 9V | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  7vPnC serotype 14 | 100.0 [90.5 to 100.0] | 100.0 [89.7 to 100.0]
  7vPnC serotype 18C | 100.0 [90.5 to 100.0] | 100.0 [90.0 to 100.0]
  7vPnC serotype 19F | 100.0 [90.0 to 100.0] | 100.0 [89.7 to 100.0]
  7vPnC serotype 23F | 97.3 [85.8 to 99.9] | 94.3 [80.8 to 99.3]
  Additional serotype 1 | 100.0 [90.5 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 3 | 100.0 [90.7 to 100.0] | 100.0 [89.7 to 100.0]
  Additional serotype 5 | 97.4 [86.2 to 99.9] | 94.1 [80.3 to 99.3]
  Additional serotype 6A | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
  Additional serotype 7F | 100.0 [90.5 to 100.0] | 100.0 [89.4 to 100.0]
  Additional serotype 19A | 100.0 [90.7 to 100.0] | 100.0 [90.0 to 100.0]
Statistical Analysis 1: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; difference in proportions = -2.6, 95% CI 2-sided [-13.9 to 8.0]
Statistical Analysis 2: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.2 to 10.6]
Statistical Analysis 3: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.4 to 10.3]
Statistical Analysis 4: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.3]
Statistical Analysis 5: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.0 to 10.1]
Statistical Analysis 6: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.1 to 10.5]
Statistical Analysis 7: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; difference in proportions = 3.0, 95% CI 2-sided [-9.1 to 16.6]
Statistical Analysis 8: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-10.0 to 10.1]
Statistical Analysis 9: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.4 to 10.3]
Statistical Analysis 10: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; difference in proportions = 3.3, 95% CI 2-sided [-8.6 to 17.2]
Statistical Analysis 11: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]
Statistical Analysis 12: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.7 to 10.6]
Statistical Analysis 13: Comparison: 7vPnC / 13vPnC vs MnCC / 13vPnC; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; difference in proportions = 0.0, 95% CI 2-sided [-9.5 to 10.0]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 4 after vaccination for local reactions and systemic events or up to Day 194 (Visit 6 / Days 166 to 194 Follow-up Telephone Visit to assess AEs)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 subject and as nonserious in another subject, or 1 subject may have experienced both a serious and nonserious event during the study.
Groups:
- 7vPnC / 13vPnC: 13vPnC administered as a single 0.5 mL dose IM. Participants had previously received 7vPnC in study D118-P8.
  Adverse Events include Local reactions and Systemic events collected on the diary card and reported in the diary-related case report form (systematic assessment) and other Adverse Events collected on the case report form (non-systematic methods).
  Other Adverse Events N=22; Local reactions N=38; Systemic events N=38.
- MnCC / 13vPnC: 13vPnC administered as a single 0.5 mL dose IM. Participants had previously received MnCC in study D118-P8.
  Adverse Events include Local reactions and Systemic events collected on the diary card and reported in the diary-related case report form (systematic assessment) and other Adverse Events collected on the case report form (non-systematic methods).
  Other Adverse Events N=20; Local reactions N=36; Systemic events N=36.
Arm/Group | 7vPnC / 13vPnC | MnCC / 13vPnC
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/36
Other Adverse Events (participants affected / at risk) | 38/38 | 36/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 7vPnC / 13vPnC (N=38) | MnCC / 13vPnC (N=36)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Congenital flat feet (Congenital, familial and genetic disorders) | 0 | 2
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Injection site pain (General disorders) | 4 | 4
Pyrexia (General disorders) | 3 | 1
Injection site swelling (General disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 2
Pharyngitis (Infections and infestations) | 2 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Gastritis viral (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Joint sprain (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 2 | 3
Hypersomnia (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Tenderness: Any (Skin and subcutaneous tissue disorders) | 35 | 31
Tenderness: Significant (Skin and subcutaneous tissue disorders) | 4 | 7
Swelling: Any (Skin and subcutaneous tissue disorders) | 4 | 2
Swelling: Mild (Skin and subcutaneous tissue disorders) | 1 | 1
Swelling: Moderate (Skin and subcutaneous tissue disorders) | 4 | 1
Redness: Any (Skin and subcutaneous tissue disorders) | 2 | 2
Redness: Mild (Skin and subcutaneous tissue disorders) | 0 | 1
Redness: Moderate (Skin and subcutaneous tissue disorders) | 2 | 1
Fever ≥38 degrees C but ≤39 degrees C (General disorders) | 1/34 | 0/35
Decreased appetite (General disorders) | 3 | 6
Decreased appetite: Mild (General disorders) | 3 | 4
Decreased appetite: Moderate (General disorders) | 1 | 3
Irritability (General disorders) | 7 | 5
Irritability: Mild (General disorders) | 5 | 4
Irritability: Moderate (General disorders) | 2 | 2
Increased sleep (General disorders) | 10 | 12
Increased sleep: Mild (General disorders) | 6 | 9
Increased sleep: Moderate (General disorders) | 5 | 5
Increased sleep: Severe (General disorders) | 1 | 0
Decreased sleep (General disorders) | 3 | 4
Decreased sleep: Mild (General disorders) | 2 | 3
Decreased sleep: Moderate (General disorders) | 1 | 1
Rash (General disorders) | 2 | 0
Rash: Mild (General disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.